CLINICAL TRIAL: NCT01190774
Title: An Investigation Into Patients' State Anxiety Reduction Following the Administration of a Dental Anxiety Questionnaire in the Dental Treatment Setting
Brief Title: Anxiety Assessment Intervention in Dental Patients
Acronym: ANXDEN
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of St Andrews (Other)
Collaborators: University of Manchester (Other)
Responsible Party: Professor Nick Tarrier, University of Manchester
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: Denanx0103
Record Dates: First submitted 2010-08-25; First posted 2010-08-30 (Estimated); Last update posted 2010-08-30 (Estimated); Status verified 2003-07

CONDITIONS: Anxiety State
Keywords: dental anxiety; state anxiety; randomised control trial; psychological intervention
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Dentist behaviour (Experimental): Patient completes the MDAS which is handed to receptionist who then gives the information to the dentist with patient knowledge
  Interventions: Behavioral: Information to health provider without patient knowledge
- Dentist behaviour and patient expectancy (Experimental): Patient completes the MDAS and hands to the dentist
  Interventions: Behavioral: dentist behaviour and patient expectancy

INTERVENTIONS:
Behavioral: Information to health provider without patient knowledge — The intervention consists of the assessment information from the MDAS questionnaire being given to the dentist via the receptionist without the knowledge of the patient
  Arms: Dentist behaviour
Behavioral: dentist behaviour and patient expectancy — patient give information about their dental anxiety to the dentist
  Arms: Dentist behaviour and patient expectancy

SUMMARY:
Dental anxiety is a significant barrier to the acceptance of regular dental care, and has many negative consequences. A study by Dailey et al. (2002) found that providing the dentist with information of the high level of a patient's dental anxiety prior to treatment using the Modified Dental Anxiety Scale (MDAS, Humphris et al., 1995), lead to a significant reduction in state anxiety from pre- to post- dental consultation compared to a control group. The current study aimed to replicate the study by Dailey et al. (2002), and to further explore whether the reduction in state anxiety associated with the MDAS could be explained by a change in dentist behaviour on receiving it, or a change in patient expectancy about the treatment session, or both.

The design was a randomised control trial involving three groups, which aimed to manipulate possible changes in dentist behaviour and patient expectancy. In Group 1, the MDAS was left at reception, as expected by the patient. In Group 2, the dentist received the MDAS, although the patient did not expect this. In Group 3 the dentist received the MDAS and the patient did expect this. The sample (N=182) was taken from two dental access centres, and included participants obtaining a score of 19 or above, or 5 on any one item of the MDAS. Pre- and post-dental consultation measures of state anxiety were taken using the six-item short-form of the state scale of the Spielberger State-Trait Anxiety Inventory (STAI-S, Marteau & Bekker, 1992).

DETAILED DESCRIPTION:
The aim of the current study was to compare the degree of anxiety reduction in dentally anxious patients attending a Dental Access Center where the dentist did or did not receive the patients' assessment of dental anxiety.

METHODS Design of study A three group pre-and post-test design was adopted, a control group (Group1: patient completed the MDAS (Modified Dental Anxiety Scale) questionnaire and handed it to the receptionist) and the experimental group where the patient handed the MDAS to the dentist (Group 3). An additional group was included (Group 2). Patients completed the MDAS and handed it to the receptionist whereupon it was given to the dentist contrary to patient expectation. The dental staff were kept blind to the actual design of the study. The Local Research and Ethics Committee approved the study.

Test the hypothesis that patients sharing assessment information about their dental anxiety to members of the dental team has beneficial effects on their state anxiety.

Randomisation A block randomisation schedule was computer generated by University of Manchester statistician (BT). Pre-sealed opaque envelopes that contained questionnaires specific to the three groups were prepared by a colleague to minimise selection bias. All materials were pre-coded with the participant number.

Sample

Dental Access Centers provide: general dental services to those who are not registered with a NHS dentist, NHS patient charges and receipt of easily available treatment and advice (appointment not always necessary). The study was conducted at two Greater Manchester Dental Access Centers. These sites offered treatment to emergency dental patients who were more likely to become dentally anxious than regular attenders (Maggirias and Locker, 2002) . Participants were volunteers recruited, from October 2003 to April 2004.

ELIGIBILITY:
Inclusion Criteria:

* scores 19 and above on MDAS
* read and write English
* 18 years of age and above

Exclusion Criteria:

* mental illness

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 182 (Actual)
Dates: Start 2003-09; Primary Completion 2004-04 (Actual); Study Completion 2004-09 (Actual)

PRIMARY OUTCOMES:
State Anxiety | immediately after dental appointment
  Speilberger's State-Trait Anxiety Inventory, short form

SECONDARY OUTCOMES:
Discussion of dental anxiety with dentist | during appointment
  Simple 'yes' 'no' dichotomy

CONTACTS AND LOCATIONS:
Overall Officials: Gerald M Humphris, PhD, Study Director — University of St Andrews
Locations (1):
- University of Manchester, Manchester, United Kingdom